CLINICAL TRIAL: NCT03856008
Title: Investigation of Morphological Changes of Cervical Spinal Stabilization Exercise Programs Focused on Flexor and Extensor Muscles in Cervical Muscles by Magnetic Resonance Imaging in Healthy Individuals
Brief Title: Effect of Cervical Spinal Stabilization Exercise Programs by Magnetic Resonance Imaging in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Erdi Kayabınar, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-180136
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: cervical spinal stabilisation exercises; muscle cross sectional area; muscle t2 relaxation time

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercises focused on flexor muscles. (Experimental): Flexor cervical stabilization exercises will be applied.
  Interventions: Other: Exercises focused on flexor muscles
- Exercises focused on extensor muscles. (Experimental): Extensor cervical stabilization exercises will be applied.
  Interventions: Other: Exercises focused on extensor muscles
- Control. (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: Exercises focused on flexor muscles — Exercises emphasis flexor muscles.
  Arms: Exercises focused on flexor muscles.
Other: Exercises focused on extensor muscles — Exercises emphasis extensor muscles.
  Arms: Exercises focused on extensor muscles.

SUMMARY:
The aim of this study was to investigate the morphological changes in the neck muscles of cervical spinal stabilization exercises focused on flexor and extensor muscles applied to healthy individuals.

DETAILED DESCRIPTION:
In the prevention and treatment of cervical region pathologies, various exercise methods are applied in the clinic. The clinical exercises vary according to the time and severity of the pathology but also according to the pathology itself. These exercises include exercises focusing on flexor or extensor muscles. The aim of this study was to investigate the morphological changes in the neck muscles of cervical spinal stabilization exercises focused on flexor and extensor muscles applied to healthy individuals. At least 27 healthy male subjects between the age of 18-30 are planned to be included in the study. Individuals will be divided into 3 groups by simple randomization method. In one group cervical stabilization exercise program focused on the flexor muscles will be applied and the other group cervical stabilization exercise program focused on the extensor muscles will be applied for 8 weeks. Individuals in the control group will only be evaluated without exercise. In the study, by using magnetic resonance imaging (MRI) method as the main evaluation, muscle anatomical cross-sectional area and T2 relaxation time measurements will be made and morphological changes in muscles will be determined. These evaluation procedures will be performed on longus colli, sternocleidomastoid, semispinalis cervicis, multifidus and upper trapezius muscles. As additional evaluation methods, muscle strength and muscle endurance tests, normal joint motion measurements, posture evaluation and MRI measurement of cervical spine curvature will be performed. All evaluations will be performed at the beginning and at the end of these 8 weeks and the effects of the exercises applied on the muscles in the two groups will be examined.

ELIGIBILITY:
Inclusion Criteria:

* being healthy
* age between 18 to 30 years
* agree to participate in the study

Exclusion Criteria:

* to undergo any surgical procedure of the vertebral column
* inflammatory disease
* rheumatological disease
* history of malignancy
* congenital spinal cord anomaly
* congenital and/or spinal deformities
* radiculopathy
* myelopathy
* other neurological disorders
* vestibular disorders and/or trauma history

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Cervical muscles cross sectional area | Change from baseline time at the end of 8 week
  Measurement of the cross-sectional area of the examined muscles by axial mri images. The circles of the muscles will be drawn by hand and examined with a computer program.
Cervical muscle T2 relaxation time | change from baseline time at the end of 8 week
  T2 relaxation time of circled muscles will be measured with milliseconds. T2 axial and t2 mapping images will be obtained with mri.

SECONDARY OUTCOMES:
Cervical muscle strength | change from baseline score at the end of 8 week
  The strength of the cervical flexor and extensor muscles and deltoid muscles will be measured by a digital hand dynamometer (Lafayette Instrument Company, USA). The measurements of the dynamometer will be based on fine muscle test positions described by Lovett. When measuring the muscle strength, resistance will be given from the frontal region for flexors and over the occipital region for the cervical extensors. Resistance for deltoid muscles will be given around the shoulder. The tests will be repeated three times and the highest of 3 repeated results obtained from these measurements will be recorded. The strength of the muscles around the scapula will be evaluated with manual muscle test, which is rated at 0-5 points developed by Lovett. 5 point is maximum and 0 is the minimum point. Statistical analyzes will be done with total muscle strength values. A total of eight muscle muscle tests will be performed to evaluate the scapular muscles.
New York posture rating chart | change from baseline score at the end of 8 week
  This evaluation system is scored by monitoring the posture changes that may occur in 13 different parts of the body. Accordingly, if the person's posture is correct five points will be given.If impairment is moderate, three points will be given and if the impairment is severe, 0 point will be given.
Tragus angle measurement | change from baseline score at the end of 8 week
  The evaluation of the tragus angle will be used as a result of the evaluation of the photograph taken in front of the checkered back surface with the computer program. The Tragus, ear and C7 vertebrae will be marked and measured.
Cervical flexor and extensor endurance test | change from baseline score at the end of 8 week
  The endurance evaluation of the deep cervical flexor muscles patients will be lied in the supine position, while the hands are in the free position on the abdomen, and the patient will be asked to remove the head slightly with the instruction. A slight amount (30%) craniocervical flexion will be required after this position has been taught to the patient. The time in which the patient maintains the position while maintaining the craniocervical flexion will be recorded in seconds. In the evaluation of endurance of deep cervical extensor muscles, the individual will be asked to lie down from T6 level and the head and neck will droop from the bed. The person will be instructed to bear the weight (4 kg in men) attached to a velcro placed over the ears in this position. The test will begin with a slight amount of craniocervical flexion, as if the individual makes head up against weight, and the time the individual maintains this position will be measured in seconds.
Cervical range of motion measurement | change from baseline score at the end of 8 week
  The Cervical Range of Motion (Performance Attainment Associates, St. Paul, MN, 55117, United States) (CROM 3) device will be used for the active evaluation of cervical range of motion. Flexion-extension, rotation and lateral flexion measurements will be performed at appropriate positions. The value found on the compass of the device will be recorded after each measurement.
Evaluation of cervical spine curvature | change from baseline score at the end of 8 week
  In the evaluation of cervical spine curvature, measurements of Cobb angle will be used on images taken in sagittal plane with MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Erdi Kayabınar, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Sıhhıye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No